CLINICAL TRIAL: NCT05508581
Title: Microwaves Ablation of Varicose Veins
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, joseph samy youssef saleeb, Principal investigator, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Microwaves ablation
Record Dates: First submitted 2021-10-22; First posted 2022-08-19 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Varicose Veins
MeSH Terms: conditions — Varicose Veins

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Varicose veins (Other): Ablation of varicose veins by microwaves
  Interventions: Procedure: microwaves ablation of varicose veins

INTERVENTIONS:
Procedure: microwaves ablation of varicose veins — Microwave ablation is an endovenous treatment. This is a similar treatment approach as laser ablation and radiofrequency ablation. "Endovenous" means that the treatment device is inside the vein during treatment.

SUMMARY:
Lower-limb varicose veins (VVs) are the most common of vascular diseases and affect up to one-third of the population, severely affecting the quality of life (QoL) of patients. In past decades, traditional surgical ligation and stripping were the gold standard therapy for patients with VVs; however, traditional methods have demonstrated high complication and recurrence rates. Thus, the practices are moving toward minimally invasive alternatives.

DETAILED DESCRIPTION:
Lower-limb varicose veins (VVs) are the most common of vascular diseases and affect up to one-third of the population, severely affecting the quality of life (QoL) of patients. In past decades, traditional surgical ligation and stripping were the gold standard therapy for patients with VVs; however, traditional methods have demonstrated high complication and recurrence rates. Thus, the practices are moving toward minimally invasive alternatives. Endo venous thermal ablation, such as radiofrequency ablation and endo venous laser ablation (EVLA), has become the recommended first-line treatment for VVs worldwide. These endo venous procedures provide a quicker recovery time and improved QoL and produce fewer complications than traditional surgery .Endo venous microwaves ablation is a minimally invasive procedure in treatment of V.V, investigators confirmed that endo venous microwave ablation (EMA) was an effective new technique for the treatment of VVs. On previous trials confirmed that the endo venous microwave ablation procedure demonstrated a shorter procedure time, lower complication, and local recurrence than the endo venous laser ablation procedure. The aim of the study was to determine whether endo venous microwave ablation of varicose vein was associated with better effectiveness and less complications and evaluate the outcome of patients who underwent endo venous microwave ablation (EMA).

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 60 years, either sex, elective admission
2. primary symptomatic VVS (CEAP,C3-C6)
3. Recurrent Varicose Veins after surgery
4. Greater saphenous vein diameter up to 3 cm
5. Greater saphenous vein with variable depth even with depth less than 6mm
6. Greater saphenous vein with tortuosity
7. Diabetic patient with risk of wound infection after surgery
8. Patient with hostile groin
9. Availability of patients for all follow-up visits

Exclusion Criteria:

1. secondary Varicose Veins
2. Acute thrombosis near the Saphenous-femoral junction
3. Recanalized Greater saphenous vein
4. pregnancy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2023-12-15 (Actual)

PRIMARY OUTCOMES:
1.Number of Participants with Lack of flow or closed great saphenous vein | 6 months
  Complete ablation of varicose veins done or if any residual remind
2.Operation time | Intraoperative
  The time of the whole procedure

SECONDARY OUTCOMES:
1. Number of Participants with recurrence varicose vein varicose veins reappear again after the operation | 12 month
  Reopening of the Varicose veins
2. Number of Participants with adverse effect of the procedure | 12 months
  Thrombophlebitis,Infection or blood loss

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Gamal glal, Lecturer, Study Chair — Lecturer at Vascular and endovascular surgery department Assuit University
Locations (1):
- Asyut University Hospitals, Faculty of Medicine, Department of Vascular Surgery .Timeframe of the study: 2 years, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No